CLINICAL TRIAL: NCT03711669
Title: Identification of Biomarkers That Help to Predict Success of Immunosuppression Withdrawal in Patients With Type 1 Autoimmune Hepatitis
Brief Title: Biomarkers to Predict the Success of Immunosuppression Withdrawal in Autoimmune Hepatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Maria Londoño, Senior Staff Specialist, Hospital Clinic of Barcelona
Other Study IDs: PI17/00955
Record Dates: First submitted 2018-10-04; First posted 2018-10-18 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Autoimmune Hepatitis
Keywords: autoimmune hepatitis; disease flare; treatment withdrawal
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Histological sample at inclusion. The following analysis will be performed: usual staining techniques to evaluate the presence of portal inflammation, interface hepatitis and fibrosis. Expression of group of genes involved in liver rejection (CXCL9, CXCL10, FoxP3, TK1, CD74, MMP9) will be evaluated with qPCR in RNA of the tissue samples cryopreserved at -80ºC. Immunochemical staining to quantity the number of lymphocytes CD4+, CD8+ and Tregs.
  * Blood samples collected at the inclusion and in every follow-up visit:
    * Frequency and characteristics of Tregs (CD4+, CD25+, CD127- and FoxP3). Intracellular stain of CTLA-4 will be evaluated as well
    * Stimulation with IL2 to study Tregs response.
  * Faecal sample at inclusion to evaluate microbiome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Immunosuppression withdrawal — IS will be tapered gradually over a period of 6 months. Azathioprine will be stopped during the first 3 months, reducing the dose 50% every month. Prednisone will be tapered 2.5mg monthly until total withdrawal. During withdrawal and the first year after stopping treatment patients will undergo laboratory tests on a monthly basis, afterwards follow-up will be done every 3 months until the end of the project.

SUMMARY:
Autoimmune hepatitis (AIH) is an inflammatory, chronic and recurrent liver disease of unknown etiology that can lead to cirrhosis or acute liver failure. It is a rare disease affecting 16 cases every 100,000 persons in Europe, mainly in women in every age group. It is characteristic the presence of high levels of aminotransferases, hypergammaglobulinemia and high titres of autoantibodies, as well as interface hepatitis in the biopsy.

Due to the autoimmune etiology of AIH, treatment is based on immunosuppressive strategies, mainly prednisone and azathioprine regimens which make possible to achieve remission in approximately 75% of cases with moderate or severe hepatocellular inflammation.

Remission is defined as a normalization in aminotransferases, immunoglobulin G (IgG) and resolution histological inflammation (this last one comes after biochemical remission). It has also been observed that there is a restoration in number and function of Tregs after achieving remission.

The rates of recurrence after withdrawing it varies from 30-87% depending on the studies and their follow-up. It is usual to maintain treatment indefinitely in clinical practice. This strategy implies maintaining treatment for long periods of time in patients that could be available to maintain sustained remission, exposing them to adverse effects. From all these, we think it is important to be able to identify patients who will be able to maintain biochemical and histological remission without immunosuppression (IS), which still is not known in this disease's management.

Some observational and retrospective studies have identified some parameters that could imply a higher risk of recurrence after stopping treatment such as high levels of aminotransferases and IgG, less time of remission before withdrawal (specifically less than 2 years) or presence of interface hepatitis in a biopsy prior discontinuation of treatment. However, the accuracy of these parameters is low and as a result, management of this disease has not changed much over the past decades, still having patients under prolonged treatment unnecessarily.

For the previously mentioned reasons, there is a need to identify new biomarkers that allow clinicians selecting patients with AIH in whom treatment could be stopped avoiding its costs and adverse effects. At the same time, it would help to understand the immunopathogenesis of AIH and identification of new therapeutic targets.

DETAILED DESCRIPTION:
Study design: This is a prospective not controlled, not randomized, unicentric study to establish predictive biomarkers for a safe and effective treatment withdrawal in patients with type 1 AIH.

Length of the study: Screening is expected to take a year. Treatment withdrawal will be done gradually over a period of 6 months and there will be a follow-up of 18 months.

Sample size: The rate of recurrence has been around 36% in some studies. However, this rate is uncertain and it depends on the studied population and the afterwards follow-up. That is why investigators have calculated the sample size with the confidence interval of this rate and a 10% precision which was of 87 patients. Expecting 10% of losses, the final sample size is 96 patients.

Patients: Investigators will select 96 patients diagnosed with type 1 AIH with biochemical remission of at least 3 years that are under immunosuppressive treatment followed in Hospital Clinic Barcelona. Patients with type 2 AIH are excluded because of their proved high risk of recurrence. Other inclusion and exclusion criteria are the following:

Treatment withdrawal: IS will be tapered gradually over a period of 6 months. Azathioprine will be stopped during the first 3 months, reducing the dose 50% every month. Prednisone will be tapered 2.5mg monthly until total withdrawal. During withdrawal and the first year after stopping treatment patients will undergo laboratory tests on a monthly basis, afterwards, follow-up will be done every 3 months until the end of the project.

Sustained remission: Patients that after stopping treatment maintain AST/ALT under 2 times the upper normal limit.

Recurrence: Patients who do not fulfil previous criteria.

Data collection:

* Demographic variables: age, sex, time from diagnosis to treatment withdrawal, laboratory information such as aminotransferases, gamma-glutamyl transferase (GGT), alkaline phosphatase (AP) and autoantibodies.
* Histological sample at the moment of inclusion in which the following analysis will be performed: usual staining techniques to evaluate the presence of portal inflammation, interface hepatitis and fibrosis. Expression of a group of genes involved in liver rejection (CXCL9, CXCL10, FoxP3, TK1, CD74, MMP9) will be evaluated with quantitative polymerase chain reaction (qPCR) in RNA of the tissue samples cryopreserved at -80ºC. Immunochemical staining to quantify the number of lymphocytes CD4+, CD8+ and Tregs.
* The following variables will be evaluated in blood samples collected at the inclusion and in every follow-up visit:

  * Flux cytometry: Frequency and characteristics of Tregs (CD4+, CD25+, CD127- and FoxP3). The intracellular stain of CTLA-4 will be evaluated as well.
  * Stimulation with interleukin 2 (IL2) to study Tregs response (measured by the expression of pSTAT5 after 20minutes of stimulation and the afterwards production of IL10).
  * Autoantibodies titers: antinuclear autoantibodies (ANA), anti-smooth muscle antibody(ASMA), anti-liver kidney microsome type 1 (antiLKM), anti-soluble liver antigen (antiSLA) and immunoglobulins levels.

Statistical analysis: Categorical variables will be compared with Chi or Fisher tests. Quantitative variables will be analyzed with non-parametric tests (Mann-Whitney for independent samples and Wilcoxon for paired samples). To quantify the expression of genes in blood and tissue sample the Ct of the gene will be normalized with the 3 "housekeeping" (18S, HPRT, GAPDH) to generate the delta Ct. Results will be expressed as a relative expression of the cDNA of the study and the calibrated sample. Differences of <0.05 will be considered as statistically significant. Data analysis will be performed with Stata vs 15.1.

Ambition: Investigator's hypothesis is that those patients affected with type 1 AIH able to maintain remission after treatment withdrawal will express distinctive serological and histological biomarkers, making possible the identification of patients that could benefit from stopping treatment in the future avoiding its costs and adverse effects. At the same time, it would help to understand the immunopathogenesis of AIH and the identification of new therapeutic targets. Therefore, changing the natural history of this disease where there has been little advance in this field in the past decades.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 AIH.
* AST/ALT within normal limits the 3 years prior inclusion.
* normal levels of IgG.
* > 18 years-old.

Exclusion Criteria:

* Presence of biochemical alterations during the 3 years prior diagnosis.
* Coexistence of another autoimmune disease that requires IS.
* Prednisone doses over 7.5mg/day.
* Biopsy prior starting withdrawal with a Knodell score over 3/16.
* Positivity for hepatitis B virus, hepatitis C virus or human immunodeficiency virus.
* Pregnancy.
* Glomerular filtrate <35ml/min.
* Not being able to attend follow-up visits.
* Use of drugs or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with type 1 AIH with biochemical remission of at least 3 years that are under immunosuppressive treatment followed in Hospital Clinic Barcelona. Patients with type 2 AIH are excluded because of their proved high risk of recurrence.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Remission rate after treatment withdrawal | Through study completion (average 1.5 years)
  Patients that after stopping treatment maintain aspartate aminotransferase (AST) and alanine aminotransferase (ALT) under 2 times the upper normal limit at the end of the study

SECONDARY OUTCOMES:
Adverse outcomes after treatment withdrawal (descriptive) | Through study completion (average 1.5 years)
  Evaluation of complications that take place after treatment withdrawal: need of hospitalization if there is a flare or diagnosis of 'de novo' autoimmune diseases or worsening symptoms such as asthenia or arthralgias.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Londoño, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital del Mar, Barcelona

IPD SHARING:
Plan to Share IPD: No
IPD are to be shared with researchers participating in the study.